CLINICAL TRIAL: NCT06986486
Title: Neoadjuvant Chemotherapy and Stereotactic Body Radiation Therapy Followed by Liver Transplantation for Unresectable Perihilar Cholangiocarcinoma: pCOLA
Brief Title: Liver Transplantation for Unresectable Perihilar Cholangiocarcinoma
Acronym: pCOLA
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 254-24
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Perihilar Cholangiocarcinoma; Klatskin Tumor
Keywords: liver transplantation; stereotactic body radiation therapy; downstaging
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and transplant specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplant: Patients with liver-limited unresectable perihilar cholangiocarcinoma with no other non-oncological contraindication to liver transplantation

SUMMARY:
This is multicentric, single-arm, observational, investigator-drive study investigating the efficacy of liver transplantation after successful downstaging/disease control of unresectable perihilar cholangiocarcinoma using chemotherapy +/- immunotherapy and stereotactic body radiation therapy (SBRT).

DETAILED DESCRIPTION:
Patients with unresectable pCCA who fit within inclusion criteria will be enrolled in the study. They will undergo staging laparoscopy with nodal sampling at the hepatic hilum. In case of negative staging (no peritoneal carcinomatosis, no positive hilar lymph nodes, negative peritoneal washing), they will receive downstaging with gemcitabine-cisplatin +/- durvalumab for 2 cycles, followed by SBRT, followed by at least 4 other cycles of gemcitabine-cisplatin +/- durvalumab. After downstaging, they will undergo disease restaging and, if at least disease stability is confirmed, they will undergo transplant screening and listing. Treatment with gemcitabine-cisplatin + durvalumab will continue until liver transplant, progression or unacceptable toxicity.

During listing, restaging will be performed every two months with CT scan and/or MRI, molecular markers and FDG-PET. The target interval between listing and transplant should be less than 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unresectable peripheral cholangiocarcinoma arising one centimeter or more above the superior pancreatic margin, with tumor diameter ≤ 3 cm, diagnosed by:
* Transcatheter biopsy or brush cytology
* CA-19.9 > 100 mg/ml and/or a mass on cross-sectional imaging with a malignant appearing stricture on cholangiography
* Biliary ploidy by FISH with a malignant appearing stricture on cholangiography
* Age between 18 years and 70 years
* Absence of intra- and extrahepatic metastases
* Absence of lymph-nodal metastases at any site
* Biliary stenting of all liver districts
* No contraindications to liver transplantation
* No concomitant malignancies or history of other malignancies in the previous 5 years
* Written informed consent

Exclusion Criteria:

* Intrahepatic cholangiocarcinoma
* Uncontrolled infection
* Concomitant malignancies or history of other malignancies in the previous 5 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver-limited unresectable perihilar cholangiocarcinoma with no other non-oncological contraindication to liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | 3 years
  To evaluate overall survival at 36 months in patients with unresectable hilar cholangiocarcinoma treated with neoadjuvant chemotherapy and SBRT followed by liver transplantation according to the modified Mayo Clinic protocol

SECONDARY OUTCOMES:
3-year recurrence-free survival | 3 years
  To evaluate recurrence-free survival at 36 months in patients with unresectable hilar cholangiocarcinoma treated with neoadjuvant chemotherapy and SBRT followed by liver transplantation according to the modified Mayo Clinic protocol
Safety and feasibility | 3 years
  To evaluate the safety and feasibility of neoadjuvant SBRT and chemotherapy in patients with unresectable hilar cholangiocarcinoma candidate to liver transplantation, in particular we will describe in detail the therapeutic path of all patients with unresectable pCCA that enter within the downstaging pathway and are evaluated for LT, how many are able to be transplanted within this protocol, and what are the reasons for dropout from the protocol
Quality of life | 3 years
  To evaluate the impact of this treatment strategy and of LT on quality of life in patients with unresectable pCCA. Quality of life will be assessed with validated questionnaires. Questionnaires will be performed at baseline and at 6 months intervals; they will be matched and compared with that of eligible patients recruited within the same study period and receiving non-transplant treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori di Milano, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: Undecided